CLINICAL TRIAL: NCT03195465
Title: The Effect of High Antioxidant Cacao on Behaviors in Children With Autism Spectrum Disorder
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution. Efforts made to contact PI unsuccessful. No study data available.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5170206
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2021-05-13 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cacao group (Experimental): 1 group of subjects will all receive the high antioxidant cacao bars. 4 squares of the dark chocolate will be administered twice daily between the hours of 6 a.m. and 6 p.m.
  Interventions: Dietary Supplement: Dark Chocolate

INTERVENTIONS:
Dietary Supplement: Dark Chocolate — Dark Chocolate bars with 70% cacao and 30% organic cane sugar where 4 squares of the dark chocolate will be administered twice daily between the hours of 6 a.m. and 6 p.m. daily for four weeks.

SUMMARY:
The purpose of this study is to determine if routine consumption of high antioxidant cacao can have an effect on the behaviors of children with Autism Spectrum Disorder. This is proposed as children with Autism Spectrum Disorder have elevated oxidative stress markers, such as, free radicals making them highly vulnerable to oxidative damage. Thus, it is proposed that foods high in antioxidant activity can offer protection against oxidative stress and thus impact behaviors.

DETAILED DESCRIPTION:
Subjects will include both males and females with an age range between 5 and 18 years. Study will include subjects from any race or ethnicity that meet eligibility criteria. Inclusion criteria: children with a diagnosis of Autism Spectrum Disorder, are between the ages of 5 and 18, and like 70% dark chocolate. Exclusion criteria: Food allergies, Caffeine hypersensitivity, Theobromine hypersensitivity, History of seizures or epilepsy, Developmental age < 24 months, and Diabetics. The target study population is school aged children with a diagnosis of Autism Spectrum Disorder. Participants will be recruited using snowballing and judgmental sampling via word-of-mouth, flyers, emails, and social media with a $50.00 gift card offered for participants who complete the study in full and $15.00 gift card for teachers who complete study in full. Flyers will be distributed throughout the Southern California area due to proximity, however, participants may come from any region if satisfying inclusion criteria and time commitment. Flyers will be placed in, but not limited to, common public places such as local community centers, pediatric therapy clinics, pediatricians' offices, churches, schools, and more. The principal student researcher or appropriate PhD committee personnel will acquire email addresses of potential participants. Specific social media outlets will include postings on, but not limited to, Facebook, Instagram, and Twitter. The name of the principal investigator and contact information of the student researcher will be available on the flyer with an invitation to contact researchers with any questions about the study. Families of those children with a diagnosis of Autism Spectrum Disorder will be offered a flyer to determine if they are interested in participating in the study. The informed consent process will be facilitated by the student researcher with the parents of the child with a diagnosis of Autism Spectrum Disorder. The informed consent process will take place at a location of convenience for parents who will be provided fifteen minutes for decision making and discussion. Due to the subjects' impaired decision making capacity, the parents will provide consent on their behalf. HIPPA compliance forms will be included with informed consent process. Privacy of medical and research records will be secured in a locked cabinet in a locked office.Procedures are listed as follows:

1. Informed Consent and HIPPA documents.
2. Subject will also be offered a taste testing of the chocolate bar to be used in the study as liking the 70% dark chocolate is part of inclusion criteria.
3. After consent is provided, parent will fill out the Youth & Adolescent Food Frequency Questionnaire based on their child's typical dietary habits, an Autism Spectrum Rating Scale, an Aberrant Behavior Checklist, and the Parental Stress Index Questionnaire.
4. Student researcher will prepare doses (4 squares per dose or 8 grams) of the dark chocolate for each child in one week increments at a time. The dark chocolate will be wrapped in foil to protect against light and kept in a sealed Ziploc bag to prevent against oxidation in order to maintain the cacao's integrity.
5. Student researcher will meet with each parent/family once per week to collect any questionnaires and to deliver the dark chocolate doses for the subsequent weeks.
6. Student researcher will meet with teachers at baseline, end of week two, and end of week four to collect all questionnaires.
7. Subject will consume 4 squares of the dark chocolate twice daily between the hours of 6 a.m. and 6 p.m.
8. Student researcher will contact parents and teachers weekly via phone/email to follow up on administration of the chocolate.
9. Parent and primary school teacher will fill out the Autism Spectrum Rating Scale and the Aberrant Behavior Checklist at the end of week two and at the end of week four.
10. Parent will fill out the Parental Stress Index Questionnaire at the end of week four.

Research analysis plan will include non-parametric statistics. For the pre-test and post-test analysis of the Parental Stress Index scale Friedman's test will be used. For all other repeated measures such as the Aberrant Behavior Checklist and the Autism Spectrum Rating Scale the Wilcoxon Signed Rank Test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Children with a diagnosis of Autism Spectrum Disorder, are between the ages of 4 and 18, and like 70% dark chocolate.

Exclusion Criteria:

* Food allergies, Caffeine hypersensitivity, Theobromine hypersensitivity, History of seizures or epilepsy, Developmental age < 24 months, and Diabetics.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Berk, DrPH, Study Chair — Loma Linda University
Locations (1):
- Loma Linda University Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Damodaran LP, Arumugam G. Urinary oxidative stress markers in children with autism. Redox Rep. 2011;16(5):216-22. doi: 10.1179/1351000211Y.0000000012. PMID 22005342
- [Background] Hardan AY, Fung LK, Libove RA, Obukhanych TV, Nair S, Herzenberg LA, Frazier TW, Tirouvanziam R. A randomized controlled pilot trial of oral N-acetylcysteine in children with autism. Biol Psychiatry. 2012 Jun 1;71(11):956-61. doi: 10.1016/j.biopsych.2012.01.014. Epub 2012 Feb 18. PMID 22342106
- [Background] Scholey AB, French SJ, Morris PJ, Kennedy DO, Milne AL, Haskell CF. Consumption of cocoa flavanols results in acute improvements in mood and cognitive performance during sustained mental effort. J Psychopharmacol. 2010 Oct;24(10):1505-14. doi: 10.1177/0269881109106923. Epub 2009 Nov 26. PMID 19942640

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cacao Group
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: PI left institution without completing results. All efforts to contact PI for data have been unsuccessful. No data available to report.
Arm/Group | Cacao Group
Number analyzed (Participants) | 0
Age, Continuous [unit: years]
Sex: Female, Male
Race (NIH/OMB)
Abberant Behavior Checklist — PI left institution. Efforts made to contact PI unsuccessful. No study data available.

OUTCOME MEASURES:

1. Primary Outcome: Aberrant Behavior Checklist 2nd Edition
Description: This is a valid and reliable tool that is made up of 58 questions comprised of 5 main content areas: Irritability; Social Withdrawal; Stereotypic Behavior, Hyperactivity Non Compliance, and Inappropriate Speech.
Time Frame: Change in subscale scores over the four weeks.
Population: PI left institution without completing results. Multiple attempts made to contact PI without success. Not data available to submit.
Arm/Group | Cacao Group
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: PI left institution without completing results. All efforts to contact PI for data have been unsuccessful. No time frame available to report.
Description: PI left institution without completing results. All efforts to contact PI for data have been unsuccessful. No data available to report.
Arm/Group | Cacao Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT03195465/Prot_SAP_000.pdf